CLINICAL TRIAL: NCT03857282
Title: The Effect of Tai Chi Exercises on Physical Activity and Pulmonary Function In Patients With Coronary Artery Bypass Grafting
Brief Title: Tai Chi Exercises on Physical Activity and Pulmonary Function in CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Maria Razzaq
Record Dates: First submitted 2019-02-08; First posted 2019-02-27 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
Keywords: Bicycling; Coronary Artery Disease; Pulmonary Function; Tai Chi
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercises (Active Comparator): Bicycling Exercise (lower Limb)
  Interventions: Other: Aerobic Exercises
- Tai Chi Exercises (Experimental): Tai Chi Exercises (yang 24 Postures)
  Interventions: Other: Tai Chi Exercises

INTERVENTIONS:
Other: Aerobic Exercises — 5 to 10 min warm up exercises than 30min bicycle exercise and 5 to 10 min cool down exercises
  Arms: Aerobic Exercises
Other: Tai Chi Exercises — 5 to 10 min warm up exercises and 30 min Tai Chi exercises and than than 5 to 10 min cool down exercises.
  Arms: Tai Chi Exercises

SUMMARY:
To improve the cardiopulmonary endurance in Coronary artery bypass grafting (CABG) patients. Internationally in cardiac hospital facility of cardiac rehabilitation is available to improve the patient's physical activity and decrease the list of secondary complications. But in Pakistan ideal phase II cardiac rehabilitation is limited available in limited hospitals due to cost issues and limited resources for monitoring during exercise. A Randomized control trail Study was conducted in Armed force institute of cardiology (AFIC) Rawalpindi. The Total sample size was 74 post (CABG). The aim of study was to influence of Tai chai on coronary artery bypass surgery patients.

DETAILED DESCRIPTION:
Coronary blood vessel disease is a disease of vessels supplying the muscles of the heart. Heart attack is generally acute condition and mainly produced by an obstruction, that stop the blood supply to the heart. Coronary artery diseases can be progressive or non-progressive. Physical activity or exercise is necessary for all the healthy individuals to prevent the risk of diseases and maintained health status. Physical exercise often varies from physical activity by animation more measured in relations of intensity and period, while physical activity studies tend to integrate an enormous diversity of unspecified activities. Physical activity or exercise is used as conservative treatment of coronary artery diseases as a cardiac rehabilitation. Cardiac rehabilitation gives positive effect on patient's conditions by the exercise training program. Exercise may improve the maximal oxygen consumption (VO2 max) and repetitive capacity or capability to maintain physical activity for long periods of time. Exercise have multiple benefits on improving endothelial function, myocardial stream replacement decreasing smoking, body mass, plasma fats and blood pressure. Guided work out or exercise may decrease the development of coronary atherosclerosis. Different types of Aerobic exercises are the part of cardiac rehabilitation, start at very early in patients with coronary artery bypass grafting. Aerobic exercises may improve the maintenance of functional capacity and muscular strength but it shows no impact on pulmonary function and respiratory muscle strength. Aerobic exercises are perform in different ways some of them are in the form of intervals and some are continues. Studies shows that Four weeks of intense training increased VO2 peak significantly after both aerobic interval training and moderate continues training, but After 6 months only aerobic interval training gives high peak oxygen uptake (VO2 peak). It shows that both training have similarly effects in the tiny tenure and in extensive tenure only effect aerobic interval training.

The most common aerobic exercises are perform at Treadmill and bicycle in cardiac rehabilitation program. Studies shows that Treadmill aerobic working out progresses both functional mobility and circulatory appropriateness in patients with chronic (CABG) and is more operational than reference rehabilitation reciprocated to conventional care. Now a day Tai chi is used in all over the world for health and defense or protection. Tai chi is a fighting art it is used in defense and health related fitness it is appropriate conditioning exercise for elder people. In health related benefits Yang Tai chi are most commonly practiced worldwide. Tai chi exercises are also practiced in rehabilitation department to gain the balance, coordination, endurance and physical activity in patients with stroke and coronary artery bypass grafting most commonly.

Consistent aerobic workout and lifestyle modification are imperative for preventing and treating high blood pressure. For individuals with hypertension

,The American College of Sports Medicine recommends the following exercise guidelines like frequency: aerobic exercise most preferably all days of a week; resistance exercise 2-3 days per week. Intensity of exercise must be moderate intensity aerobic and resistance exercise. Time of exercise must be 30-60 minutes for every day of aerobic implementation while resistance working out at least one set of 8-12 reiterations for each of the main muscle groups. Studies shows that Tai Chi gives positive effects on blood pressure. Tai Chi training may reduce the systolic and diastolic blood pressure in patients with HTN. Tai chi also reduce the systolic as well as diastolic in normal healthy individuals.

Young DR, conducted a study with the title of "The properties of aerobic workout and Tai Chi on blood pressure in older individuals" and they concluded that the programs of low and modest concentration workout have the same effects on blood pressure in elderly patients.

Stroke is a common root of expiry in ageing population it is due to atherosclerosis are hemorrhagic in the minor or intermediate vessels of the brain. In such kind of patient significant reduction in quality of life, neurological discrepancies and deficiency of intellectual function.It reported that stroke patients increasing peak oxygen acceptance and walking distance by workout. Cerebrovascular accident patients frequently have compromised equilibrium and motor function, thus Tai Chi training program can be used in rehabilitation of stroke. A study in elderly subjects on Tai chi, balancing exercise and workout instruction groups. After four months of physical activity the follow up evaluation illustrate that only Tai Chi subjects informed that their daily activities and their whole life had been exaggerated. The result demonstrates that in women emotional as well as physical control is supposed to be improved in sense of enhancement in overall well-being and inspiration to continue physical training also rises.

Effectiveness of Tai Chi, brisk hiking, meditation and reading in reducing psychological and emotional stress in 1992 and calculated that Tai Chi activities are used to decrease mental stress or disorder it is advantageous to quit smoking, drinking and other life threatening obsessions also. For the reason that Tai Chi is also used as to enlarge psychological well being and mental sickness.

Another study concluded that Tai Chi trainings are an aerobic movements it is very supportive for different age and gender, it also increase functional capability of the participants.

There was a research gap in previous study Tai chi training was done after phase II cardiac rehabilitation and duration of training was 6 months to 1 year. In current study we analyze Effect of Tai chi exercise on physical activity, pulmonary function and the rate of perceived exertion after exercise in patients with cardiovascular bypass surgeries in phase II cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* post-operative CABG patients,
* Ejection fraction >40% were included

Exclusion Criteria:

* 2,3,4 scale of angina,
* unstable congestive heart failure,
* Substantial myocardial ischemia,
* Cardiac arrhythmias,
* Reopen chest after surgery,
* Uncontrolled diabetes and hypertension

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
forced expiratory volume in one second (FEV1) | 6 weeks
  Changes from the Baseline, forced expiratory volume in one second (FEV1) in liters will be measured through Digital spirometer
Forced vital capacity (FVC) | 6 weeks
  Changes from the Baseline, forced vital capacity (FVC) in liters will be measured through Digital spirometer
Peak expiratory flow (PEF). | 6 weeks
  Changes from the Baseline, Peak expiratory flow (PEF) in Liters/seconds will be measured through Digital spirometer
International physical activity questionnaire (IPAQ) | 6 weeks
  Changes from Baseline, (IPAQ) It is recommended that activity bouts of greater than 3 hours are truncated. That is to say that a bout cannot be longer than 3 hours (180 minutes). This means that in each category a maximum of 21 hours of activity are permitted a week (3 hours X 7 days) To calculate metabolic equivalent (MET) minutes a week multiply the MET value given (remember walking = 3.3, moderate activity = 4, vigorous activity = 8) by the minutes the activity was carried out and again by the number of days that that activity was undertaken. For example if someone reports walking for 30 minutes 5 days a week then the total MET minutes for that activity are 3.3 X 30 X 5=495 Met minutes a week.
  You can add the MET minutes achieved in each category (walking, moderate activity and vigorous activity) to get total MET minutes of physical activity a week.

SECONDARY OUTCOMES:
Modified Borg's rating of perceived exertion (RPE) scale | 6 weeks
  (RPE) Scale - Modified BORG scale. Grading scale for fatigue and endurance. 0. At rest. 1. Very easy. 2. Somewhat easy. 3. Moderate. 4. Somewhat hard. 5. Hard 7 very Hard and 10 very, very hard
Heart Rate | 6 weeks
  Changes from the Baseline; Heart Rate (beats per minute)
Oxygen Saturation (SPO2) | 6 weeks
  Changes from the Baseline; Saturation in Percentage
Blood Pressure | 6 weeks
  Changes from the Baseline; Blood Pressure in (mmHg)
Heart Rate Reserve | 6 weeks
  Changes from the Baseline; Heart Rate Reserve beat per minute
Respiratory Rate | 6 weeks
  Changes from the Baseline; Respiratory Rate breath per minute

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid Baig, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith SC Jr, Collins A, Ferrari R, Holmes DR Jr, Logstrup S, McGhie DV, Ralston J, Sacco RL, Stam H, Taubert K, Wood DA, Zoghbi WA. Our time: a call to save preventable death from cardiovascular disease (heart disease and stroke). Circulation. 2012 Dec 4;126(23):2769-75. doi: 10.1161/CIR.0b013e318267e99f. Epub 2012 Sep 17. No abstract available. PMID 22988010
- [Background] Bergheanu SC, Bodde MC, Jukema JW. Pathophysiology and treatment of atherosclerosis : Current view and future perspective on lipoprotein modification treatment. Neth Heart J. 2017 Apr;25(4):231-242. doi: 10.1007/s12471-017-0959-2. PMID 28194698
- [Background] Stary HC, Chandler AB, Glagov S, Guyton JR, Insull W Jr, Rosenfeld ME, Schaffer SA, Schwartz CJ, Wagner WD, Wissler RW. A definition of initial, fatty streak, and intermediate lesions of atherosclerosis. A report from the Committee on Vascular Lesions of the Council on Arteriosclerosis, American Heart Association. Circulation. 1994 May;89(5):2462-78. doi: 10.1161/01.cir.89.5.2462. PMID 8181179
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults--United States, 2006. MMWR Morb Mortal Wkly Rep. 2007 Nov 9;56(44):1157-61. PMID 17989644
- [Background] Edwards DG, Schofield RS, Lennon SL, Pierce GL, Nichols WW, Braith RW. Effect of exercise training on endothelial function in men with coronary artery disease. Am J Cardiol. 2004 Mar 1;93(5):617-20. doi: 10.1016/j.amjcard.2003.11.032. PMID 14996592
- [Background] Gielen S, Hambrecht R. Effects of exercise training on vascular function and myocardial perfusion. Cardiol Clin. 2001 Aug;19(3):357-68. doi: 10.1016/s0733-8651(05)70222-8. PMID 11570110
- [Background] Villella M, Villella A. Exercise and cardiovascular diseases. Kidney Blood Press Res. 2014;39(2-3):147-53. doi: 10.1159/000355790. Epub 2014 Jul 29. PMID 25117881
- [Background] Pattyn N, Beckers PJ, Cornelissen VA, Coeckelberghs E, De Maeyer C, Frederix G, Goetschalckx K, Possemiers N, Schepers D, Van Craenenbroeck EM, Wuyts K, Conraads VM, Vanhees L. The effect of aerobic interval training and continuous training on exercise capacity and its determinants. Acta Cardiol. 2017 Jun;72(3):328-340. doi: 10.1080/00015385.2017.1304712. Epub 2017 Mar 21. PMID 28636505
- [Background] Macko RF, Ivey FM, Forrester LW, Hanley D, Sorkin JD, Katzel LI, Silver KH, Goldberg AP. Treadmill exercise rehabilitation improves ambulatory function and cardiovascular fitness in patients with chronic stroke: a randomized, controlled trial. Stroke. 2005 Oct;36(10):2206-11. doi: 10.1161/01.STR.0000181076.91805.89. Epub 2005 Sep 8. PMID 16151035
- [Background] Hollings M, Mavros Y, Freeston J, Fiatarone Singh M. The effect of progressive resistance training on aerobic fitness and strength in adults with coronary heart disease: A systematic review and meta-analysis of randomised controlled trials. Eur J Prev Cardiol. 2017 Aug;24(12):1242-1259. doi: 10.1177/2047487317713329. Epub 2017 Jun 5. PMID 28578612